CLINICAL TRIAL: NCT02071862
Title: Ph1 Study of the Safety, PK, and PDn of Escalating Oral Doses of the Glutaminase Inhibitor CB-839, as a Single Agent and in Combination With Standard Chemotherapy in Patients With Advanced and/or Treatment-Refractory Solid Tumors
Brief Title: Study of the Glutaminase Inhibitor CB-839 in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CX-839-001
Record Dates: First submitted 2014-02-14; First posted 2014-02-26 (Estimated); Last update posted 2022-07-20 (Actual); Status verified 2020-02

CONDITIONS: Solid Tumors; Triple-Negative Breast Cancer; Non Small Cell Lung Cancer; Renal Cell Carcinoma; Mesothelioma; Fumarate Hydratase (FH)-Deficient Tumors; Succinate Dehydrogenase (SDH)-Deficient Gastrointestinal Stromal Tumors (GIST); Succinate Dehydrogenase (SDH)-Deficient Non-gastrointestinal Stromal Tumors; Tumors Harboring Isocitrate Dehydrogenase-1 (IDH1) and IDH2 Mutations; Tumors Harboring Amplifications in the cMyc Gene
Keywords: Tumor metabolism; Glutaminase; Glutamine; Tricarboxylic acid (TCA) cycle
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Mesothelioma | interventions — CB-839; Paclitaxel; Everolimus; Docetaxel; cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- CB-839 (Experimental): CB-839 administered as oral capsules two (BID) or three times daily (TID) in 21-day cycles until disease progression or unacceptable toxicity
  Interventions: Drug: CB-839
- Pac-CB (Experimental): CB-839 administered as oral capsules twice daily (BID) in combination with standard dose paclitaxel in 28-day cycles until disease progression or unacceptable toxicity
  Interventions: Drug: CB-839; Drug: Pac-CB
- CBE (Experimental): CB-839 administered as oral capsules twice daily (BID) in combination with standard dose everolimus in 28-day cycles until disease progression or unacceptable toxicity
  Interventions: Drug: CB-839; Drug: CBE
- CB-Erl (Experimental): CB-839 administered as oral capsules twice daily (BID) in combination with standard dose erlotnib in 28-day cycles until disease progression or unacceptable toxicity
  Interventions: Drug: CB-839; Drug: CB-Erl
- CBD (Experimental): CB-839 administered as oral capsules twice daily (BID) in combination with standard dose docetaxel in 21-day cycles until disease progression or unacceptable toxicity
  Interventions: Drug: CB-839; Drug: CBD
- CB-Cabo (Experimental): CB-839 administered as oral capsules twice daily (BID) in combination with standard dose cabozantinib in 28-day cycles until disease progression or unacceptable toxicity
  Interventions: Drug: CB-Cabo

INTERVENTIONS:
Drug: CB-839 — CB-839 monotherapy
  Other Names: Glutaminase Inhibitor
  Arms: CB-839; CB-Erl; CBD; CBE; Pac-CB
Drug: Pac-CB — CB-839 in combination with standard dose paclitaxel
  Other Names: combo CB-839 and Paclitaxel
  Arms: Pac-CB
Drug: CBE — CB-839 in combination with standard dose everolimus
  Other Names: combo CB-839 and everolimus
  Arms: CBE
Drug: CB-Erl — CB-839 in combination with standard dose erlotnib
  Other Names: combo CB-839 and erlotnib
  Arms: CB-Erl
Drug: CBD — CB-839 in combination with standard dose docetaxel
  Other Names: combo CB-839 and docetaxel
  Arms: CBD
Drug: CB-Cabo — CB-839 in combination with standard dose cabozantinib
  Other Names: combo CB-839 and cabozantinib
  Arms: CB-Cabo

SUMMARY:
Many tumor cells, in contrast to normal cells, have been shown to require the amino acid glutamine to produce energy for growth and survival. To exploit the dependence of tumors on glutamine, CB-839, a potent and selective inhibitor of the first enzyme in glutamine utilization, glutaminase, will be tested in this Phase 1 study in patients with solid tumors.

This study is an open-label Phase 1 evaluation of CB-839 in patients with advanced solid tumors. The study will be conducted in 2 parts. Part 1 is a dose escalation study enrolling patients with locally-advanced, metastatic and/or refractory solid tumors to receive CB-839 capsules orally twice or three times daily.

In Part 2, patients with each of the following diseases will be enrolled: A) Triple-Negative Breast Cancer, B) Non-Small Cell Lung Cancer (adenocarcinoma), C) Renal Cell Cancer, D) Mesothelioma, E) Fumarate hydratase (FH)-deficient tumors, F) Succinate dehydrogenase (SDH)-deficient gastrointestinal stromal tumors (GIST), G) SDH-deficient non-GIST tumors, H) tumors harboring mutations in isocitrate dehydrogenase-1 (IDH1) or IDH2, and I) cMyc mutation tumors.

As an extension of Parts 1 & 2, patients will be treated with CB-839 in combination with standard chemotherapy. Combination groups include: Pac-CB, CBE, CB-Erl, CBD, and CB-Cabo. Pac-CB: patients with locally-advanced or metastatic TNBC will be treated with paclitaxel and CB-839. CBE: patients with advanced clear cell RCC or papillary RCC will be treated with everolimus in combination with CB-839. CB-Erl: patients with advanced NSCLC lacking the T790M EGFR mutation will be treated with erlotinib and CB-839. CBD: patients with NSCLC harboring KRAS mutation will be treated with docetaxel and CB-839. CB-Cabo: patients with histologically confirmed diagnosis of locally-advanced, inoperable or metastatic RCC treated with cabozantinib in combination with CB-839.

All patients will be assessed for safety, pharmacokinetics (plasma concentration of drug), pharmacodynamics (inhibition of glutaminase), biomarkers (biochemical markers that may predict responsiveness in later studies), and tumor response.

ELIGIBILITY:
Inclusion criteria

* Advanced malignancy that is relapsed and/or refractory to all available therapies that will confer clinical benefit. Newly diagnosed patients who refuse standard treatment regimens are also eligible
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
* Life Expectancy of at least 3 months
* Adequate hepatic, renal, cardiac, and hematologic function
* Measurable disease by RECIST criteria
* Ability to provide written informed consent in accordance with federal, local, and institutional guidelines

Exclusion Criteria

* Any other current or previous malignancy
* Chemotherapy, radiation therapy, hormonal therapy, immunotherapy or biological therapy, or investigational agent within 21 days
* Unable to receive medications oral medications
* Major surgery within 28 days before Cycle 1 Day 1
* Active infection requiring within 2 weeks prior to first dose of study drug
* Patients who have HIV, Hepatitis A, B or C or CMV reactivation
* Significant neurotoxicity/neuropathy (Grade 3 or higher) within 14 days of first dose of study drug
* Conditions that could interfere with treatment or protocol-related procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2014-02; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of CB-839: Incidence of adverse events | Every 21 days from study start until disease progression or unacceptable toxicity, assessed for an expected average of 6 months

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the Curve (AUC) of CB-839 concentration in blood | Study Days 1, 15, and 22
Pharmacodynamics: % inhibition of glutaminase in blood | Study Days 1 and 15
Clinical activity: Change in tumor volume from baseline | Every 9 weeks until disease progression or unacceptable toxicity, assessed for an expected average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Whiting, MD, PhD, Study Director — Calithera Biosciences, Inc
Locations (13):
- United States (13):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Florida Cancer Specialists, Sarasota, Florida
  - Winship Cancer Institute of Emory School of Medicine, Atlanta, Georgia
  - NIH - NCI - Center for Cancer Research, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas